CLINICAL TRIAL: NCT04692844
Title: The Mechanism of Tremor Modulating Properties of Propranolol and Primidone in Essential Tremor: A Study With Transcranial Magnetic Stimulation and Eye Blink Classical Conditioning Paradigm
Brief Title: Pathophysiology of Tremor-modulating Mechanisms of Propranolol and Primidone in Essential Tremor
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Kojović, doc. dr. Maja Kojović, dr. med., University Medical Centre Ljubljana
Other Study IDs: 0120-525/2017
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Essential Tremor
Keywords: Essential tremor; Primidone; Propranolol
MeSH Terms: conditions — Essential Tremor | interventions — Propranolol; Primidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with essential tremor treated with Propranolol: Patients will be recruited from the outpatient clinic for extrapyramidal disorders. Only patients with the diagnosis of ET made according to the newest consensus statement on the classification of tremors and only patients who will receive Propranolol in the course of routine medical practice, will be included.
  Interventions: Drug: Propranolol
- Patients with essential tremor treated with Primidone: Patients will be recruited from the outpatient clinic for extrapyramidal disorders. Only patients with the diagnosis of ET made according to the newest consensus statement on the classification of tremors and only patients who will receive Primidone in the course of routine medical practice, will be included.
  Interventions: Drug: Primidone

INTERVENTIONS:
Drug: Propranolol — Patients will receive Propranolol in the course of their routine treatment. Results will be used to explore biological phenomena or disease processes.
  Groups: Patients with essential tremor treated with Propranolol
Drug: Primidone — Patients will receive Primidone in the course of their routine treatment. Results will be used to explore biological phenomena or disease processes.
  Groups: Patients with essential tremor treated with Primidone

SUMMARY:
Pathophysiology of tremor-modulating mechanisms of propranolol and primidone in essential tremor (ET) will be studied using accelerometry with electromyography (EMG), transcranial magnetic stimulation (TMS), and eyeblink conditioning paradigm (EBCC). TMS is a well-established experimental method for studying the effects of drugs on motor cortex excitability. EBCC is a learning paradigm that can be used for studying cerebellar dysfunction since only brainstem and cerebellar functions seem to be needed for this paradigm. The investigators will use TMS to study the mechanisms of primidone and propranolol action in ET, EBCC paradigm to evaluate cerebellar dysfunction in ET patients and to show whether cerebellar dysfunction influences the effectiveness of propranolol and primidone. The investigators will clinically assess patients using The Essential Tremor Rating Assessment Scale (TETRAS) and the Scale for the Assessment and Rating of Ataxia (SARA) scales. Patients with ET will be studied prior to treatment with propranolol or primidone and re-tested 3-6 months after treatment initiation. On each visit, the investigators will clinically assess the patients and perform accelerometry, TMS measurements, and the eyeblink classical conditioning (EBCC) paradigm. The investigators hypothesize that in ET patients, baseline electrophysiological parameters will differ between responders and non-responders to propranolol and primidone and that propranolol and primidone will cause a different pattern of change in electrophysiological parameters among responders. It is hypothesized that cerebellar dysfunction will negatively correlate with patients' response to treatment.

DETAILED DESCRIPTION:
Background: Although ET is the most common of movement disorders, its pathophysiology has not yet been fully explained. Central nervous system functional studies have shown that oscillatory activity within the cerebello-thalamo-cortical networks plays a key role in ET's pathophysiology. The origin of this oscillatory activity and the potential role of the primary motor cortex in its formation or modulation remains unknown. Neuropathological studies found degenerative structural changes in the cerebellum of ET patients. Propranolol and primidone are the first-line therapies for ET and the sole medications for treating ET with the level A recommendations according to the latest guidelines of the American Academy of Neurology. Propranolol is a beta-blocker class of medication and primidone is a barbiturate. In spite of solid evidence of their effectiveness in ET patients, the mechanisms of their central action are not yet fully understood. It is believed that propranolol mediates its therapeutic action through peripheral beta-2 adrenergic receptors of skeletal muscles and muscle spindles and through central beta-adrenergic and serotoninergic receptors. After oral intake, primidone is partially metabolized to phenylethylmalonamide (PEMA) and phenobarbital. Even though the studies have shown that PEMA does not have anti-tremor activity, primidone is much more effective in alleviating tremor than phenobarbital alone. In addition, it has been shown that the anti-tremor effect of primidone occurs sooner than its metabolite phenobarbital is produced. This may be due to the non-metabolized primidone compound having an anti-tremor activity or due to PEMA's and phenobarbital's synergistic activity. No association between anti-tremor activity and the concentration of primidone or phenobarbital in the serum has been found. While phenobarbital activity is well known to be mediated through binding to gamma-aminobutyric acid (GABA) A receptors, the mechanism of action of non-metabolized primidone is poorly understood.

Aims: To study the mechanisms of primidone and propranolol action in ET with the use of TMS. The investigators believe that studying mechanisms of action of medications that have been shown to reduce ET can further improve the understanding of ET pathophysiology. Since the cerebellum is thought to be involved in ET pathophysiology the EBCC paradigm will be used to evaluate cerebellar dysfunction in ET patients and to show whether cerebellar dysfunction influences the effectiveness of propranolol and primidone.

Patients and inclusion/exclusion criteria: Fifty patients will be recruited from the outpatient clinic for extrapyramidal disorders. Only patients with the diagnosis of ET made according to the newest consensus statement on the classification of tremors and only patients who will be initiated on propranolol or primidone will be included. Exclusion criteria for TMS will be used. Patients having a history of seizures or mental illness, patients with a cardiac pacemaker, metal material in the head (except dental material in the mouth), or with medication pumps and pregnant women will be excluded from the study.

Study protocol: Patients treated with propranolol or primidone will be studied prior to treatment and 3 - 6 months after treatment initiation. Patients will not be allowed to start any new medication with the action on the central nervous system, while included in the study. Tremor will be assessed clinically using the TETRAS scale and by EMG and accelerometry recordings. Positive treatment response will be defined as a 30% or more decrease in tremor amplitude. At baseline cerebellar function will be assessed clinically with the SARA scale and electrophysiologically using the EBCC paradigm. TMS will be used to study motor cortex excitability.

Methods:

Accelerometry with electromyography: Tremor (frequency and amplitude) will be objectively evaluated in the subjects with accelerometry. A triaxial accelerometer will be attached to the 3rd metacarpal bone bilaterally. Simultaneously EMG will be recorded. Bipolar Ag / AgCl surface EMG electrodes will be placed over the flexor carpi radialis and the extensor carpi radialis muscle bilaterally. Electromyography and accelerometry will be recorded while subjects will be sitting in an armchair/wheelchair or lying in a hospital bed (a) at rest position (b) with arms outstretched (postural condition) (c) at the postural condition with 500 g mass attached to the hand (weight loading) and (d) while performing a goal-directed task (action).

Transcranial magnetic stimulation (TMS) Single TMS pulses will be applied using Magstim 2002 magnetic stimulator with monophasic waveform (Magstim Company, Carmarthenshire, Wales, UK). For double TMS pulses, two Magstim 2002 stimulators connected with the Bistim module will be used. The stimulators will be connected to a standard figure 8 coil. The coil will be positioned tangentially to the skull and over the 'hotspot' point on the scalp, with the handle pointing backward at an angle of ~ 45 ° with respect to the sagittal plane. Hotspot point is defined as stimulation site resulting in the largest motor evoked potentials (MEPs) recorded over the contralateral abductor pollicis brevis (APB) muscle. A hotspot point will be found by visual inspection. The MEP amplitude in APB muscle will be measured with EMG.

The eyeblink classical conditioning (EBCC) paradigm is a protocol of associative motor learning in which paired presentation of a conditioned (CS) and unconditioned stimulus (US) leads to the production of a conditioned eyeblink response (CR) 10,42. The CS will be a tone with a frequency of 2000 Hz and a strength of 50-70 dB higher than the hearing threshold of the subject (but at least 80 dB) and a duration of 400 milliseconds that will be presented bilaterally via binaural headphones. The unconditioned stimulus will be delivered by percutaneous supraorbital nerve electrical stimulation through a pair of Ag-AgCl cup electrodes with the cathode over the supraorbital foramen and the anode 2 cm above. Percutaneous electrical stimulation of the supraorbital nerve will last 200 microseconds and will start 200 microseconds before the end of the CS so that the stimuli will co-terminate. Blinking will be recorded with EMG electrodes placed bilaterally over the orbicularis oculi muscles. The test will consist of seven sets. In the first six sets, there will be nine trials with paired conditioned-unconditioned stimuli, one trial with the only US, and one trial with only CS. In the seventh section, eleven trials of only CS will be given. Among the individual tests, there will be a random interval (from 10s to 30s), so that the habituation will be as small as possible.

Statistical analysis: Clinical and TMS measures before and after treatment will be compared using parametric or nonparametric two-related-samples T-test, depending on the data distribution or repeated-measures ANOVA. Regression analyses will be used to determine demographic, clinical, and electrophysiological predictors of response to treatment.

It is hypothesized by investigators that in ET patients, baseline electrophysiological parameters will differ between patients who will improve while taking propranolol or primidone (responders) and patients who will not improve while taking any of these medications (non-responders). Propranolol and primidone will cause a different pattern of change in electrophysiological parameters among responders. Since the intention component of action tremor usually responds to treatment to a lesser degree than other components of tremor and is reported to be associated with cerebellar dysfunction, the investigators hypothesize that cerebellar dysfunction will negatively correlate with the patient's response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of essential tremor made according to the newest consensus statement on the classification of tremors
* patients initiated on propranolol or primidone

Exclusion Criteria:

* a history of seizures
* a history of mental illness,
* having a cardiac pacemaker
* having metal material in the head (except dental material in the mouth)
* having a medication pump
* pregnancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the outpatient clinic for extrapyramidal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Electrophysiological correlations of clinical effect | 3-6 months
  Comparison of TMS and clinical measures before and after treatment, comparison of cerebellar dysfunction with response to treatment
Effect of cerebellar function assessed by eye blink classical conditioning on drug effectiveness | 3-6 months
  Comparison of cerebellar function of responders and non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Maja Kojović, PhD, MD, Principal Investigator — maja.kojovic@kclj.si
Locations (1):
- Departmet of Neurology, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deuschl G, Raethjen J, Lindemann M, Krack P. The pathophysiology of tremor. Muscle Nerve. 2001 Jun;24(6):716-35. doi: 10.1002/mus.1063. PMID 11360255
- [Background] Kapogiannis D, Wassermann EM. Transcranial magnetic stimulation in Clinical Pharmacology. Cent Nerv Syst Agents Med Chem. 2008 Dec;8(4):234-240. doi: 10.2174/187152408786848076. PMID 19122782
- [Background] Kuo SH, Erickson-Davis C, Gillman A, Faust PL, Vonsattel JP, Louis ED. Increased number of heterotopic Purkinje cells in essential tremor. J Neurol Neurosurg Psychiatry. 2011 Sep;82(9):1038-40. doi: 10.1136/jnnp.2010.213330. Epub 2010 Aug 27. PMID 20802031
- [Background] Zesiewicz TA, Elble RJ, Louis ED, Gronseth GS, Ondo WG, Dewey RB Jr, Okun MS, Sullivan KL, Weiner WJ. Evidence-based guideline update: treatment of essential tremor: report of the Quality Standards subcommittee of the American Academy of Neurology. Neurology. 2011 Nov 8;77(19):1752-5. doi: 10.1212/WNL.0b013e318236f0fd. Epub 2011 Oct 19. PMID 22013182
- [Background] Guan XM, Peroutka SJ. Basic mechanisms of action of drugs used in the treatment of essential tremor. Clin Neuropharmacol. 1990 Jun;13(3):210-23. doi: 10.1097/00002826-199006000-00003. No abstract available. PMID 1972653
- [Background] Buijink AW, van der Stouwe AM, Broersma M, Sharifi S, Groot PF, Speelman JD, Maurits NM, van Rootselaar AF. Motor network disruption in essential tremor: a functional and effective connectivity study. Brain. 2015 Oct;138(Pt 10):2934-47. doi: 10.1093/brain/awv225. Epub 2015 Aug 5. PMID 26248468
- [Background] Ziemann U, Lonnecker S, Steinhoff BJ, Paulus W. Effects of antiepileptic drugs on motor cortex excitability in humans: a transcranial magnetic stimulation study. Ann Neurol. 1996 Sep;40(3):367-78. doi: 10.1002/ana.410400306. PMID 8797526
- [Background] Kronenbuerger M, Gerwig M, Brol B, Block F, Timmann D. Eyeblink conditioning is impaired in subjects with essential tremor. Brain. 2007 Jun;130(Pt 6):1538-51. doi: 10.1093/brain/awm081. Epub 2007 Apr 27. PMID 17468116
- [Background] Ghassemi NH, Marxreiter F, Pasluosta CF, Kugler P, Schlachetzki J, Schramm A, Eskofier BM, Klucken J. Combined accelerometer and EMG analysis to differentiate essential tremor from Parkinson's disease. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:672-675. doi: 10.1109/EMBC.2016.7590791. PMID 28268417
- [Background] Hopfner F, Haubenberger D, Galpern WR, Gwinn K, Van't Veer A, White S, Bhatia K, Adler CH, Eidelberg D, Ondo W, Stebbins GT, Tanner CM, Helmich RC, Lenz FA, Sillitoe RV, Vaillancourt D, Vitek JL, Louis ED, Shill HA, Frosch MP, Foroud T, Kuhlenbaumer G, Singleton A, Testa CM, Hallett M, Elble R, Deuschl G. Knowledge gaps and research recommendations for essential tremor. Parkinsonism Relat Disord. 2016 Dec;33:27-35. doi: 10.1016/j.parkreldis.2016.10.002. Epub 2016 Oct 4. PMID 27769649
- [Background] Louis ED, Faust PL, Vonsattel JP, Honig LS, Rajput A, Robinson CA, Rajput A, Pahwa R, Lyons KE, Ross GW, Borden S, Moskowitz CB, Lawton A, Hernandez N. Neuropathological changes in essential tremor: 33 cases compared with 21 controls. Brain. 2007 Dec;130(Pt 12):3297-307. doi: 10.1093/brain/awm266. Epub 2007 Nov 19. PMID 18025031
- [Background] Hedera P, Cibulcik F, Davis TL. Pharmacotherapy of essential tremor. J Cent Nerv Syst Dis. 2013 Dec 22;5:43-55. doi: 10.4137/JCNSD.S6561. PMID 24385718
- [Background] Calzetti S, Findley LJ, Pisani F, Richens A. Phenylethylmalonamide in essential tremor. A double-blind controlled study. J Neurol Neurosurg Psychiatry. 1981 Oct;44(10):932-4. doi: 10.1136/jnnp.44.10.932. PMID 7031184
- [Background] Ondo W. Essential Tremor: What We Can Learn from Current Pharmacotherapy. Tremor Other Hyperkinet Mov (N Y). 2016 Mar 4;6:356. doi: 10.7916/D8K35TC3. eCollection 2016. PMID 26989572
- [Background] Clark RE, Manns JR, Squire LR. Trace and delay eyeblink conditioning: contrasting phenomena of declarative and nondeclarative memory. Psychol Sci. 2001 Jul;12(4):304-8. doi: 10.1111/1467-9280.00356. PMID 11476097